CLINICAL TRIAL: NCT04687033
Title: The Effect of The Ten-Session Dual-tDCS On Lower-Limb Performance in Sub- Acute and Chronic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: MU-CIRB 2019
Record Dates: First submitted 2020-12-09; First posted 2020-12-29 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Stroke, Ischemic
MeSH Terms: conditions — Ischemic Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dual-tDCS & PT (Experimental): Dual tDCS: the anodal tDCS will be applied over the M1 of the lesioned hemisphere, while the cathodal tDCS will be applied over the M1 of the non-lesioned hemisphere for 20 mins before physical therapy (about
  1 hour). The current intensity is fixed at 2 mA and the current will flow continuously. Physical therapist will give an intervention program for lower limb performance.
  Interventions: Device: Transcranial direct current stimulation
- Sham-tDCS & PT (Active Comparator): Sham tDCS: the anodal tDCS will be applied over the M1 of the lesioned hemisphere, while the cathodal tDCS will be applied over the M1 of the non-lesioned hemisphere, the current intensity will be 2mA (sham mode). Physical therapist will give an intervention program for lower limb performance.
  Interventions: Device: Transcranial direct current stimulation

INTERVENTIONS:
Device: Transcranial direct current stimulation — This instrument will be used to induce post-stroke motor recovery, two different monocephalic montages are typically used to restore excitability in the lesioned hemisphere and to down-regulate excitability of the non-lesioned hemisphere and rebalance Interhemispheric inhibition. each participant will undergo a 20-minute period of tDCS, applied at 2 mA through a pair of saline-soaked surface sponge electrodes (35 cm2).

SUMMARY:
The present study aims to determine the effect of the ten-session dual tDCS combine with physical therapy on gait performance, balance, and lower limbs muscle strength in patients with subacute and chronic stroke.

DETAILED DESCRIPTION:
Stroke is a leading cause of long-term disability. The recovery of motor function after stroke is often incomplete, despite classical rehabilitation techniques. At the beginning of the 21st century, transcranial direct current stimulation (tDCS) was introduced as a non-invasive tool to reversibly modulate brain excitability in humans in which a device sends constant low direct current (DC) delivered to the area of interest through the electrodes. Transcranial direct current stimulation (tDCS) has been used in neurorehabilitation to benefit ischemic stroke patients at a different stage of stroke especially during acute, sub-acute and chronic phase with positive and safety reports.

After stroke, the excitability of the lesioned hemisphere is decreased and seen like overactive of the excitability of the non-lesioned hemisphere. Abnormally high interhemispheric inhibition (IHI) drive from intact to lesioned hemisphere has been reported. The neural plasticity begins in the early stages after stroke. Prevent the imbalance IHI and increase the excitability of the lesioned hemisphere in the early phase would be beneficial for stroke rehabilitation.

Based on the polarity-specific effects, anodal tDCS increases cortical excitability and cathodal tDCS decreases cortical excitability. Transcranial direct current stimulation (tDCS) can be applied in two distinct montages: monocephalic and bi-hemispheric/dual-tDCS (applying two electrodes over both cerebral hemispheres at the same time). To induce post-stroke motor recovery, two different monocephalic montages are typically used: i) to restore excitability in the lesioned hemisphere: anode over the lesioned hemisphere and the cathode as the reference electrode placed over the contra-orbital area ii) to down-regulate the excitability of the non-lesioned hemisphere and rebalance IHI: cathode over the non-lesioned hemisphere and the anode as the reference electrode. Dual-tDCS can be also applied, permitting simultaneous coupling of excitatory and inhibitory effects on both cortices. Few evidences are showing that tDCS (monocephalic and bi-hemispheric/dual-tDCS) could improve lower limb performance at immediate and at least 3 months. However, there is still unclear effect on gait performance and muscle strength.

Recently, dual-hemisphere tDCS which excites one hemisphere using anodal stimulation and inhibits the other by cathodal stimulation has been described in healthy volunteers to greater enhance hand motor learning compared to uni-hemispheric tDCS. The corresponding tDCS-induced changes were reported in imaging study to involve interhemispheric interactions. Dual tDCS has been more recently used in rehabilitation aiming to reduce the inhibition exerted by the non-lesioned hemisphere on the lesioned hemisphere and restore the normal balance of the IHI. Dual-tDCS combined with training or simultaneous occupational/physical therapy has been reported to improve motor skill learning and functions of the paretic upper limb in chronic stroke patients.

Lower-limb functions are commonly disabling after stroke, however, few studies have focused on the effect of tDCS on lower limb functions. A single session of anodal tDCS over the lower limb M1 has been reported to acutely enhance the effect of motor practice of the paretic ankle, force production of the paretic knee extensors, and postural stability in chronic stroke patients. A study showed an improvement in walking speed immediately after a single session of dual-tDCS alone in sub-acute stroke patients.

Based on the previous study, 1-2 mA current intensity of tDCS is usually used for modulating brain activity. The proper current density delivered is between 0.029-0.008 mA/cm 2. The higher current density, the longer-lasting, stronger, and deeper cortical neuron stimulation. Therefore, 2 mA current intensity of tDCS was applied in stroke patients for lower limb performance improvement. Following homologous brain regions, the motor area of lower extremities is in depth and previous studies demonstrated that current intensity 2 mA of tDCS could pass through the lower extremities area of the brain.

Moreover, Tahtis et al, 2013 found that using 2 mA of dual-tDCS could improve walking speed immediately after a single session in sub-acute stroke and Klomjai et al, 2018 found that a single session of dual-tDCS 2 mA with physical therapy in sub-acute stroke immediately improved sit to stand performance greater than physical therapy alone. The mechanisms of action were hypothesized that when stimulation continuously affects neuronal plasticity changes. Therefore, they suggested that further study shall implement more sessions of dual-tDCS combined with physical therapy to improve lower limb performance and determine the long lasting-after effect.

A previous study reported that the 10-consecutive sessions of tDCS were an effective treatment strategy in reducing the risk of falls and improving lower limb functions after a stroke. However, gait ability and lower limb muscle strength were not included in the outcome measures. In this study, the long-lasting effect was demonstrated at least one week to three months. There are evidences that 10 sessions for uni-hemisphere tDCS appeared to improve lower limb motor functions without serious adverse effects in patients with stroke. It is still unclear the effect of multiple sessions of dual-tDCS on gait performance and muscle strength as well as the long-lasting after-effect of multiple sessions of dual-tDCS.

Therefore, the present study aims to investigate the efficacy of ten sessions of dual-tDCS combined with conventional physical therapy on the lower limb functions after stroke in sub-acute. Clinical outcomes for lower limb performance evaluations will consist of muscle strength assessed by hand-held dynamometer, the Time up and go test for lower limb functional performance, Five times sit to stand test for dynamic balance and muscle strength, and the Zebris Force distribution measurement (FDM) for gait analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age range 20-75 years
* First ever-ischemic lesion in the territory of middle cerebral artery or anterior cerebral artery. Diagnostic confirmation will be performed by CT scan or MRI
* Sub-acute onset (1-6 months after the stroke onset) or Chronic (6 months - 5 years)
* Able to walk without physical assistance at least 6 meters

Exclusion Criteria:

* Not cooperative or cannot understand the instruction
* Clinical unstable such as vital sign unstable (systolic blood pressure (SBP) ≥ 185 mmHg or diastolic blood pressure (DBP) ≥ 110 mmHg (98) and resting heart rate averaging ≥ 100 bpm (99))
* No clear neurological antecedent history or psychiatric disorder
* Moderate pain in any joint of both lower limb (Pain Scale (VAS) ≥ 4/10)
* Unstable medical conditions such as being in the middle of changing medical treatment.
* Condition that may increase the risk of stimulation such as epilepsy, pregnancy, unexplained headaches, intracranial metal, pacemaker (evaluating by subjective examination).
* Participate in the other protocol or receive alternative treatment such as transcranial magnetic stimulation within 1 month.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline gait speed at post-intervention | immediately post-intervention
  Force distribution measurement (FDM; The WinFDM and platform, Zebris Medical GmbH, Germany) will be used to analyze step length in centimeters (cm).
  Participants will walk 3 meters per trial on a platform and be assessed 5 times. The result will be selected from an average of five trials. Participants can rest between trials for about 2 minutes or as long as they desired to avoid fatigue.
Change from baseline gait speed at 1 week post-intervention | 1 week post-intervention
  Force distribution measurement (FDM; The WinFDM and platform, Zebris Medical GmbH, Germany) will be used to analyze step length in centimeters (cm).
  Participants will walk 3 meters per trial on a platform and be assessed 5 times. The result will be selected from an average of five trials. Participants can rest between trials for about 2 minutes or as long as they desired to avoid fatigue.
Change from baseline gait speed at 1 month post-intervention | 1 month post-intervention
  Force distribution measurement (FDM; The WinFDM and platform, Zebris Medical GmbH, Germany) will be used to analyze step length in centimeters (cm).
  Participants will walk 3 meters per trial on a platform and be assessed 5 times. The result will be selected from an average of five trials. Participants can rest between trials for about 2 minutes or as long as they desired to avoid fatigue.
Change from baseline gait speed at 2 month post-intervention | 2 month post-intervention
  Force distribution measurement (FDM; The WinFDM and platform, Zebris Medical GmbH, Germany) will be used to analyze step length in centimeters (cm).
  Participants will walk 3 meters per trial on a platform and be assessed 5 times. The result will be selected from an average of five trials. Participants can rest between trials for about 2 minutes or as long as they desired to avoid fatigue.
Change from baseline gait speed at 3 month post-intervention | 3 month post-intervention
  Force distribution measurement (FDM; The WinFDM and platform, Zebris Medical GmbH, Germany) will be used to analyze step length in centimeters (cm).
  Participants will walk 3 meters per trial on a platform and be assessed 5 times. The result will be selected from an average of five trials. Participants can rest between trials for about 2 minutes or as long as they desired to avoid fatigue.

SECONDARY OUTCOMES:
Change from baseline spatiotemporal gait variable at post-intervention | immediately post-intervention
  Force distribution measurement (FDM; The WinFDM and platform, Zebris Medical GmbH, Germany) will be used to analyze step length in centimeters (cm).
  Participants will walk 3 meters per trial on a platform and be assessed 5 times. The result will be selected from an average of five trials. Participants can rest between trials for about 2 minutes or as long as they desired to avoid fatigue.
Change from baseline spatiotemporal gait variable at 1 week | 1 week post-intervention
  Force distribution measurement (FDM; The WinFDM and platform, Zebris Medical GmbH, Germany) will be used to analyze step length in centimeters (cm).
  Participants will walk 3 meters per trial on a platform and be assessed 5 times. The result will be selected from an average of five trials. Participants can rest between trials for about 2 minutes or as long as they desired to avoid fatigue.
Change from baseline spatiotemporal gait variable at 1 month | 1 month post-intervention
  Force distribution measurement (FDM; The WinFDM and platform, Zebris Medical GmbH, Germany) will be used to analyze step length in centimeters (cm).
  Participants will walk 3 meters per trial on a platform and be assessed 5 times. The result will be selected from an average of five trials. Participants can rest between trials for about 2 minutes or as long as they desired to avoid fatigue.
Change from baseline spatiotemporal gait variable at 2 months | 2 months post-intervention
  Force distribution measurement (FDM; The WinFDM and platform, Zebris Medical GmbH, Germany) will be used to analyze step length in centimeters (cm).
  Participants will walk 3 meters per trial on a platform and be assessed 5 times. The result will be selected from an average of five trials. Participants can rest between trials for about 2 minutes or as long as they desired to avoid fatigue.
Change from baseline spatiotemporal gait variable at 3 months | 3 months post-intervention
  Force distribution measurement (FDM; The WinFDM and platform, Zebris Medical GmbH, Germany) will be used to analyze step length in centimeters (cm).
  Participants will walk 3 meters per trial on a platform and be assessed 5 times. The result will be selected from an average of five trials. Participants can rest between trials for about 2 minutes or as long as they desired to avoid fatigue.
Change from baseline muscle strength at post-intervention | immediately post-intervention
  The hand-held dynamometer (HHD) measures the muscle strength in Newton. The HHD is simple, quantitative evaluation and widely used for measurement of muscle strength. The strength of lower limbs (hip flexor, hip extensor, hip abductor, knee flexor, knee extensor, ankle dorsiflexor and ankle plantarflexor) were assessed by using the hand-held dynamometer. The strength of lower limbs included hip flexor, hip extensor, hip abductor, knee flexor, knee extensor, ankle dorsiflexor and ankle plantarflexor were assessed by using the hand-held dynamometer. Hip flexor,ankle dorsiflexor and ankle plantarflexor was assessed in supine position, knee extensor was assessed in sitting position, hip extensor and knee flexor were assessed in prone position and hip abductor was assessed in side lying position. Each muscle was assessed 2 times and selected score of the best trial. Participants can rest between trials about 1 minute or as long as they desired to avoid fatigue.
Change from baseline muscle strength at 1 week | 1 week post-intervention
  The hand-held dynamometer (HHD) measures the muscle strength in Newton. The HHD is simple, quantitative evaluation and widely used for measurement of muscle strength. The strength of lower limbs (hip flexor, hip extensor, hip abductor, knee flexor, knee extensor, ankle dorsiflexor and ankle plantarflexor) were assessed by using the hand-held dynamometer. The strength of lower limbs included hip flexor, hip extensor, hip abductor, knee flexor, knee extensor, ankle dorsiflexor and ankle plantarflexor were assessed by using the hand-held dynamometer. Hip flexor,ankle dorsiflexor and ankle plantarflexor was assessed in supine position, knee extensor was assessed in sitting position, hip extensor and knee flexor were assessed in prone position and hip abductor was assessed in side lying position. Each muscle was assessed 2 times and selected score of the best trial. Participants can rest between trials about 1 minute or as long as they desired to avoid fatigue.
Change from baseline muscle strength at 1 month | 1 month post-intervention
  The hand-held dynamometer (HHD) measures the muscle strength in Newton. The HHD is simple, quantitative evaluation and widely used for measurement of muscle strength. The strength of lower limbs (hip flexor, hip extensor, hip abductor, knee flexor, knee extensor, ankle dorsiflexor and ankle plantarflexor) were assessed by using the hand-held dynamometer. The strength of lower limbs included hip flexor, hip extensor, hip abductor, knee flexor, knee extensor, ankle dorsiflexor and ankle plantarflexor were assessed by using the hand-held dynamometer. Hip flexor,ankle dorsiflexor and ankle plantarflexor was assessed in supine position, knee extensor was assessed in sitting position, hip extensor and knee flexor were assessed in prone position and hip abductor was assessed in side lying position. Each muscle was assessed 2 times and selected score of the best trial. Participants can rest between trials about 1 minute or as long as they desired to avoid fatigue.
Change from baseline muscle strength at 2 months | 2 months post-intervention
  The hand-held dynamometer (HHD) measures the muscle strength in Newton. The HHD is simple, quantitative evaluation and widely used for measurement of muscle strength. The strength of lower limbs (hip flexor, hip extensor, hip abductor, knee flexor, knee extensor, ankle dorsiflexor and ankle plantarflexor) were assessed by using the hand-held dynamometer. The strength of lower limbs included hip flexor, hip extensor, hip abductor, knee flexor, knee extensor, ankle dorsiflexor and ankle plantarflexor were assessed by using the hand-held dynamometer. Hip flexor,ankle dorsiflexor and ankle plantarflexor was assessed in supine position, knee extensor was assessed in sitting position, hip extensor and knee flexor were assessed in prone position and hip abductor was assessed in side lying position. Each muscle was assessed 2 times and selected score of the best trial. Participants can rest between trials about 1 minute or as long as they desired to avoid fatigue.
Change from baseline muscle strength at 3 months | 3 months post-intervention
  The hand-held dynamometer (HHD) measures the muscle strength in Newton. The HHD is simple, quantitative evaluation and widely used for measurement of muscle strength. The strength of lower limbs (hip flexor, hip extensor, hip abductor, knee flexor, knee extensor, ankle dorsiflexor and ankle plantarflexor) were assessed by using the hand-held dynamometer. The strength of lower limbs included hip flexor, hip extensor, hip abductor, knee flexor, knee extensor, ankle dorsiflexor and ankle plantarflexor were assessed by using the hand-held dynamometer. Hip flexor,ankle dorsiflexor and ankle plantarflexor was assessed in supine position, knee extensor was assessed in sitting position, hip extensor and knee flexor were assessed in prone position and hip abductor was assessed in side lying position. Each muscle was assessed 2 times and selected score of the best trial. Participants can rest between trials about 1 minute or as long as they desired to avoid fatigue.
Change from baseline FMA-LE at post-intervention | immediately post-intervention
  Fugl-Meyer Assessment Lower Extremity
Change from baseline FMA-LE at 1 week | 1 week post-intervention
  Fugl-Meyer Assessment Lower Extremity
Change from baseline FMA-LE at 1 month | 1 month post-intervention
  Fugl-Meyer Assessment Lower Extremity
Change from baseline FMA-LE at 2 months | 2 months post-intervention
  Fugl-Meyer Assessment Lower Extremity
Change from baseline FMA-LE at 3 months | 3 months post-intervention
  Fugl-Meyer Assessment Lower Extremity
Change from baseline Stroke Impact Scale at post-intervention | immediately post-intervention
  A questionnaire with good psychometric properties aims to evaluate stroke patient's quality of life after stroke incident. It composes of 59 items that aim to assesses 8 domains (i.e., the patient's strength, function of the hand, activities of daily living (ADL)/instrumental ADL (IADL), mobility, communication, emotion, memory and thinking, and participation in society. Each item will be scored from 1 to 5. Each domain's score ranges from 0 to 100. The higher scores mean the better self-report in participant's health.
Change from baseline Stroke Impact Scale at 1 week | 1 week post-intervention
  A questionnaire with good psychometric properties aims to evaluate stroke patient's quality of life after stroke incident. It composes of 59 items that aim to assesses 8 domains (i.e., the patient's strength, function of the hand, activities of daily living (ADL)/instrumental ADL (IADL), mobility, communication, emotion, memory and thinking, and participation in society. Each item will be scored from 1 to 5. Each domain's score ranges from 0 to 100. The higher scores mean the better self-report in participant's health.
Change from baseline Stroke Impact Scale at 1 month | 1 month post-intervention
  A questionnaire with good psychometric properties aims to evaluate stroke patient's quality of life after stroke incident. It composes of 59 items that aim to assesses 8 domains (i.e., the patient's strength, function of the hand, activities of daily living (ADL)/instrumental ADL (IADL), mobility, communication, emotion, memory and thinking, and participation in society. Each item will be scored from 1 to 5. Each domain's score ranges from 0 to 100. The higher scores mean the better self-report in participant's health.
Change from baseline Stroke Impact Scale at 2 months | 2 months post-intervention
  A questionnaire with good psychometric properties aims to evaluate stroke patient's quality of life after stroke incident. It composes of 59 items that aim to assesses 8 domains (i.e., the patient's strength, function of the hand, activities of daily living (ADL)/instrumental ADL (IADL), mobility, communication, emotion, memory and thinking, and participation in society. Each item will be scored from 1 to 5. Each domain's score ranges from 0 to 100. The higher scores mean the better self-report in participant's health.
Change from baseline Stroke Impact Scale at 3 months | 3 months post-intervention
  A questionnaire with good psychometric properties aims to evaluate stroke patient's quality of life after stroke incident. It composes of 59 items that aim to assesses 8 domains (i.e., the patient's strength, function of the hand, activities of daily living (ADL)/instrumental ADL (IADL), mobility, communication, emotion, memory and thinking, and participation in society. Each item will be scored from 1 to 5. Each domain's score ranges from 0 to 100. The higher scores mean the better self-report in participant's health.
Change from baseline Timed-up and go test (TUG) at post-intervention | immediately post-intervention
  The Timed-up & Go (TUG) test is a simple and quick functional mobility test that requires a subject to stand up, walk 3 m., turn, walk back, and then sit down.
  The objective of TUG is to determine fall risk and measure the progress of balance, sit to stand, and walking.
  This test was initially designed for elderly persons but is used for people with Parkinson's, stroke, Alzheimer's, CVA, Huntington's disease, and others.
  The TUG will be assessed only for 1 trial and participants will be performed at a comfortable speed. Materials of TUG are composed of a chair with armrest, stopwatch, and tape (to mark 3 meters). Participants will start in a seated position. After that, the participant will stand up upon therapist's command, walks 3 meters, turns around, walks back to the chair, and sits down. The time will stop when the participant is seated. Participants are allowed to use an assistive device during performing the task and this will be noted.
Change from baseline Timed-up and go test (TUG) at 1 week | 1 week post-intervention
  The Timed-up & Go (TUG) test is a simple and quick functional mobility test that requires a subject to stand up, walk 3 m., turn, walk back, and then sit down.
  The objective of TUG is to determine fall risk and measure the progress of balance, sit to stand, and walking.
  This test was initially designed for elderly persons but is used for people with Parkinson's, stroke, Alzheimer's, CVA, Huntington's disease, and others.
  The TUG will be assessed only for 1 trial and participants will be performed at a comfortable speed. Materials of TUG are composed of a chair with armrest, stopwatch, and tape (to mark 3 meters). Participants will start in a seated position. After that, the participant will stand up upon therapist's command, walks 3 meters, turns around, walks back to the chair, and sits down. The time will stop when the participant is seated. Participants are allowed to use an assistive device during performing the task and this will be noted.
Change from baseline Timed-up and go test (TUG) at 1 month | 1 month post-intervention
  The Timed-up & Go (TUG) test is a simple and quick functional mobility test that requires a subject to stand up, walk 3 m., turn, walk back, and then sit down.
  The objective of TUG is to determine fall risk and measure the progress of balance, sit to stand, and walking.
  This test was initially designed for elderly persons but is used for people with Parkinson's, stroke, Alzheimer's, CVA, Huntington's disease, and others.
  The TUG will be assessed only for 1 trial and participants will be performed at a comfortable speed. Materials of TUG are composed of a chair with armrest, stopwatch, and tape (to mark 3 meters). Participants will start in a seated position. After that, the participant will stand up upon therapist's command, walks 3 meters, turns around, walks back to the chair, and sits down. The time will stop when the participant is seated. Participants are allowed to use an assistive device during performing the task and this will be noted.
Change from baseline Timed-up and go test (TUG) at 2 months | 2 months post-intervention
  The Timed-up & Go (TUG) test is a simple and quick functional mobility test that requires a subject to stand up, walk 3 m., turn, walk back, and then sit down.
  The objective of TUG is to determine fall risk and measure the progress of balance, sit to stand, and walking.
  This test was initially designed for elderly persons but is used for people with Parkinson's, stroke, Alzheimer's, CVA, Huntington's disease, and others.
  The TUG will be assessed only for 1 trial and participants will be performed at a comfortable speed. Materials of TUG are composed of a chair with armrest, stopwatch, and tape (to mark 3 meters). Participants will start in a seated position. After that, the participant will stand up upon therapist's command, walks 3 meters, turns around, walks back to the chair, and sits down. The time will stop when the participant is seated. Participants are allowed to use an assistive device during performing the task and this will be noted.
Change from baseline Timed-up and go test (TUG) at 3 months | 3 months post-intervention
  The Timed-up & Go (TUG) test is a simple and quick functional mobility test that requires a subject to stand up, walk 3 m., turn, walk back, and then sit down.
  The objective of TUG is to determine fall risk and measure the progress of balance, sit to stand, and walking.
  This test was initially designed for elderly persons but is used for people with Parkinson's, stroke, Alzheimer's, CVA, Huntington's disease, and others.
  The TUG will be assessed only for 1 trial and participants will be performed at a comfortable speed. Materials of TUG are composed of a chair with armrest, stopwatch, and tape (to mark 3 meters). Participants will start in a seated position. After that, the participant will stand up upon therapist's command, walks 3 meters, turns around, walks back to the chair, and sits down. The time will stop when the participant is seated. Participants are allowed to use an assistive device during performing the task and this will be noted.
Change from baseline Five Times Sit to Stand Test (FTSTS) at post-intervention | immediately post-intervention
  The Five-Times-Sit-to-Stand test (FTSTS) measures the functional strength of the lower limbs. It is a clinical test that explores postural control and lower limbs muscular strength, devised to accommodate patients who can perform the sit-to-stand activity at least five times. As such, it is a helpful test in quantifying a daily transitional movement while also helping to assess fall risk and disability.
  Participants will sit with their arms folded across the chest and their back against the chair's backrest. They will be asked to stand up fully and sit down again 5 times as quickly as possible. The test will be repeated 2 times. Participants will be allowed to rest between trials for about 2 minutes or as long as they desire to avoid fatigue. The score will be selected from the best trial.
Change from baseline Five Times Sit to Stand Test (FTSTS) at 1 week | 1 week post-intervention
  The Five-Times-Sit-to-Stand test (FTSTS) measures the functional strength of the lower limbs. It is a clinical test that explores postural control and lower limbs muscular strength, devised to accommodate patients who can perform the sit-to-stand activity at least five times. As such, it is a helpful test in quantifying a daily transitional movement while also helping to assess fall risk and disability.
  Participants will sit with their arms folded across the chest and their back against the chair's backrest. They will be asked to stand up fully and sit down again 5 times as quickly as possible. The test will be repeated 2 times. Participants will be allowed to rest between trials for about 2 minutes or as long as they desire to avoid fatigue. The score will be selected from the best trial.
Change from baseline Five Times Sit to Stand Test (FTSTS) at 1 month | 1 month post-intervention
  The Five-Times-Sit-to-Stand test (FTSTS) measures the functional strength of the lower limbs. It is a clinical test that explores postural control and lower limbs muscular strength, devised to accommodate patients who can perform the sit-to-stand activity at least five times. As such, it is a helpful test in quantifying a daily transitional movement while also helping to assess fall risk and disability.
  Participants will sit with their arms folded across the chest and their back against the chair's backrest. They will be asked to stand up fully and sit down again 5 times as quickly as possible. The test will be repeated 2 times. Participants will be allowed to rest between trials for about 2 minutes or as long as they desire to avoid fatigue. The score will be selected from the best trial.
Change from baseline Five Times Sit to Stand Test (FTSTS) at 2 months | 2 months post-intervention
  The Five-Times-Sit-to-Stand test (FTSTS) measures the functional strength of the lower limbs. It is a clinical test that explores postural control and lower limbs muscular strength, devised to accommodate patients who can perform the sit-to-stand activity at least five times. As such, it is a helpful test in quantifying a daily transitional movement while also helping to assess fall risk and disability.
  Participants will sit with their arms folded across the chest and their back against the chair's backrest. They will be asked to stand up fully and sit down again 5 times as quickly as possible. The test will be repeated 2 times. Participants will be allowed to rest between trials for about 2 minutes or as long as they desire to avoid fatigue. The score will be selected from the best trial.
Change from baseline Five Times Sit to Stand Test (FTSTS) at 3 months | 3 months post-intervention
  The Five-Times-Sit-to-Stand test (FTSTS) measures the functional strength of the lower limbs. It is a clinical test that explores postural control and lower limbs muscular strength, devised to accommodate patients who can perform the sit-to-stand activity at least five times. As such, it is a helpful test in quantifying a daily transitional movement while also helping to assess fall risk and disability.
  Participants will sit with their arms folded across the chest and their back against the chair's backrest. They will be asked to stand up fully and sit down again 5 times as quickly as possible. The test will be repeated 2 times. Participants will be allowed to rest between trials for about 2 minutes or as long as they desire to avoid fatigue. The score will be selected from the best trial.

CONTACTS AND LOCATIONS:
Overall Officials: Wanalee Klomjai, PhD, Study Director — MU
Locations (1):
- Mahidol University, Nakhon Pathom, Thailand

IPD SHARING:
Plan to Share IPD: No